CLINICAL TRIAL: NCT00983671
Title: Optimising and Standardising Measurements of Inflammatory Markers in Exhaled Breath (EB) and Exhaled Breath Condensate (EBC)
Brief Title: Standardisation of Measurements in Exhaled Breath and Exhaled Breath Condensate.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Drs. M.D. Ottink, Fellow pediatric pulmonology, Pediatric Pulmonology, dept. of Pediatrics, University Hospital Maastricht
Other Study IDs: MEC 09-2-080; NL25969.068.09
Record Dates: First submitted 2009-09-17; First posted 2009-09-24 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Asthma; Cystic Fibrosis; Chronic Lung Disease; Pneumonia
Keywords: Asthma; cystic fibrosis; chronic lung disease; bronchopulmonary dysplasia; pneumonia
MeSH Terms: conditions — Asthma; Cystic Fibrosis; Pneumonia; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Exhaled breath condensate. Exhaled breath.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- children with asthma: children with diagnosed asthma, age 6-18 years
- cystic fibrosis: children with cystic fibrosis, age 6-18 years
- chronic lung disease: children with chronic lung disease, also known as bronchopulmonary dysplasia, age 6-18 years
- pneumonia: children with clinical signs of pneumonia, age 6-18 years

SUMMARY:
Background: in various pediatric pulmonary diseases such as asthma, cystic fibrosis or bronchopulmonary dysplasia an increased inflammation is present. Measuring this inflammation is often hardly possible and requires invasive techniques such as bronchoscopy.

With the use of exhaled breath condensate (EBC) or exhaled breath (EB) analysis it is possible to measure the inflammation in an non-invasive way. However, there is a great need to further standardise these measurements and to identify possible confounding factors.

DETAILED DESCRIPTION:
Background of the study:

Measurement of inflammatory markers (IM) in exhaled breath and exhaled breath condensate (EB(C)) is a very interesting and useful non-invasive new technique to evaluate airway inflammation. This technique is helpful for diagnostic and monitoring purposes in both children and adults with chronic lung disease. The hypothesis of the present study is that standardisation not only increase the reproducibility of measurements but will also enlarge the possibility to detect differences between healthy and diseased subjects.

Objective of the study:

1. to investigate the influence of various factors on the concentration of markers in EB(C); parameters on a subject level (e.g. breathing pattern, nose clip, inspiratory filter, saliva contamination, physical exertion), on an apparatus level (cleaning procedures, temperature of the condenser tube, environmental conditions, buffer bags), and on a measurement/analysis level (sampling time, storage time, storage temperature, protein inhibitor or bovine serum albumine) can be discriminated.
2. to assess whether the reproducibility of measurements in EB(C) can be increased by analysing with ellipsometry, lyophilization or by standardising for exhaled volume, sampling time, or dilution factor.
3. to investigate whether differences in inflammatory markers (IM) in EBC between healthy and diseased subjects will increase by specific EB(C) sampling from more distal airways. Children with asthma, cystic fibrosis (CF), primary ciliary dyskinesia (PCD), bronchopulmonary dysplasia (BPD), and lower respiratory tract infections (LRTI) will be included.

Study design:

Part I: Cross-sectional study assessing the random influence of presence or absence of various factors on the concentration of IM in EB(C); Part II: A short-term prospective study on reproducibility during five consecutive days; Part III: A cross-sectional comparative study in several groups of children (healthy, asthma, CF, PCD, BPD, LRTI);

Study population:

Study part I and II are performed in healthy adult volunteers. Study part III is performed in healthy children and in children with asthma, CF, PCD, BPD, and LRTI aged 2-16 years.

Primary study parameters/outcome of the study:

Study part I: Concentration of IM in EB(C). Study part II: Reproducibility as assessed by coefficients of variations of IM in EB(C).

Study part III: Concentration of IM in EB(C) from more distal and more proximal airways.

ELIGIBILITY:
Inclusion Criteria:

study part I and II:

* healthy adults, 18-50 years study part III:
* healthy children age 6-18 years
* patients with cystic fibrosis
* patients with asthma
* patients with chronic lung disease
* patients with pneumonia, all age 6-18 years

Exclusion Criteria:

Study part I and II:

* Subjects with a history of atopy or respiratory disease, as indicated by the ISAAC questionnaire.

Study part III:

* Mental retardation
* active smoking
* heart disease
* syndromes
* congenital malformations of the airways
* inability to perform the measurements
* for patients with lower respiratory tract infection: oxygen need, asthma or other chronic lung disease, active or passive smoking, inability to perform the measurements.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: For study I and II: community sample For study III: healthy children recruited at a primary school, children with asthma, cystic fibrosis, chronic lung disease or pneumonia, recruited from the outpatient clinic of pediatric pulmonology
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Study I: concentration of inflammatory markers in EB(C) | 1 week
Study II: Reproducibility of inflammatory markers in EB(C) | 1 week
Study III: concentration of inflammatory markers in EB(C) of the proximal and distal airways | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: E. Dompeling, PhD, Study Director — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Pediatric Pulmonology, Maastricht, Po Box 5800, Netherlands